CLINICAL TRIAL: NCT06063226
Title: Clinical and Microbiological Aspects of Probiotics in Non-surgical Periodontal Therapy: a Randomized Controlled Trial.
Brief Title: Clinical and Microbiological Aspects of Probiotics in Non-surgical Periodontal Therapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Collaborators: Probiotical S.p.A. (Industry)
Responsible Party: Principal Investigator, Prof. Marco Dolci, Full Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARO
Record Dates: First submitted 2023-09-26; First posted 2023-10-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis; Probiotics; Non Surgical Periodontal Therapy
Keywords: lactobacillus rhamnosus; lactobacillus plantarum; supportive periodontal therapy; non surgical periodontal therapy
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics (Experimental): Patients who will be assigned to oral consumption of one stick of probiotics with L. plantarum and L. rhamnosus for 30 days, in adjucntion to routinary oral hygiene procedures.
  Interventions: Other: Experimental
- Positive Control (Placebo Comparator): Patients who will be assigned to oral consumption of one stick of placebo for 30 days, in adjucntion to routinary oral hygiene procedures.
  Interventions: Other: Positive control
- Negative control (Other): Patients who will be assigned to routinary oral hygiene procedures esclusively.
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Experimental — Orally administred probiotics with L. plantarum and L. rhamnosus
  Other Names: Orally administration of probiotics with L. plantarum and L. rhamnosus
  Arms: Probiotics
Other: Negative control — Only routinary oral hygiene procedures
  Other Names: Only routinary oral hygiene procedures
  Arms: Negative control
Other: Positive control — Orally administred placebo without probiotics
  Other Names: Orally administred placebo without probiotics
  Arms: Positive Control

SUMMARY:
The goal of this randomized clinical trial is to test the effect orally administration of Probiotics based on Lactobacillus rhamnosus LR04 and Lactobacillus plantarum LP14 as adjuvant in people suffering from periodontitis stage II-III. The main questions it aims to answer are:

* QUESTION 1: orally administered probiotics based on the previous strains could represent a useful tool in support of non-surgical periodontal therapy in reducing clinical periodontal indexes?
* QUESTION 2: orally administered probiotics based on the previous strains could represent a useful tool in support of non-surgical periodontal therapy in reduce the amount of periodontal pathogens in periodontal pockets?

Partecipants in the test group will take the test probiotic for 90 days in adjunction of the routinary oral hygiene procedures.

Partecipants in the positive controlled group will take the placebo for 90 days in adjunction of the routinary oral hygiene procedures.

Partecipants in the negative control group will perform only the routinary oral hygiene procedures.

Researchers will compare 3 groups to see if orally administered probiotics based on L. rhamnosus and L. plantarum may hel in the reduction of periodontal indexes and of the periodontal pathogen bacteria.

DETAILED DESCRIPTION:
The diagnosis of periodontitis passes through the recording of periodontal probing values on 6 sites for each periodontal element, the recording of clinical indices such as the percentage of bleeding sites and those with plaque, finally through the execution of a full-x-ray consisting of intraoral films that guarantee staging through the calculation of the loss of clinical attachment, corresponding to the loss of alveolar bone caused by the disease. The therapy of periodontitis is composed of several steps and begins with the control of the biofilm. This control is carried out with professional supragingival hygiene sessions followed by subgingival instrumentation of the periodontal pockets in order to remove the hard and soft deposits below the gingival margin, which would not otherwise be eliminated with the supragingival strategy alone. The response to mechanical therapy and the risk of relapses go hand in hand with the patient's response, his ability to maintain a good level of oral hygiene at home and to keep return appointments. In this sense, dental research has worked hard to develop additional aids to mechanical therapy to try to improve its performance. In the last decade in particular, the use of probiotics has found an increasingly wider field in periodontology, as they are based on the idea of enhancing the eubiosis ratios of the non-pathogenic flora in order to make the environment unfavorable for the proliferation of a pathogenic flora.

The present study aims to evaluate whether the quarterly oral administration of probiotics based on Lactobacillus plantarum LP14 and Lactobacillus rhamnosus LR04 can improve the response to non-surgical periodontal therapy of subgingival instrumentation in patients suffering from stage II-III periodontitis and complexity of grade A-B.

Primary objective To evaluate the adjuvant effect of probiotics based on Lactobacillus plantarum LP14 and Lactobacillus rhamnosus LR04 in non-surgical periodontal therapy.

Secondary objective Characterize the microbiological picture of patients with periodontitis with and without the aid of probiotics.

MATERIALS AND METHODS Three groups of volunteers of both sexes will be enrolled for the study without age restrictions.

Inclusion criteria Patients in the absence of other systemic pathologies reported in the medical history, smokers and non-smokers, non-drinkers, in the absence of previous or current administration of other sources of probiotics, capable of providing informed consent.

Exclusion criteria Subjects with a history of systemic diseases (diabetes, autoimmune diseases, inflammatory bowel diseases, neurodegenerative diseases), drinkers, who take or have taken probiotics in the last 3 months, unable to provide informed consent.

Minimum sample size Sample size calculation (Alpha = 0.05; Power = 95%) for 3 independent study groups, and a continuous primary endpoint. Sample size = Z2 (1-alpha/2) p (1-p) / d2 Where Z(1-alpha/2) is the standard variate corresponding to 1.96 at 5% type 1 error, p is the expected proportion in the population expressed in decimals based on previous studies and d is the confidence level decided by the researcher expressed in decimal. Regarding the primary outcome of Bleeding On Probing (BOP), the expected difference between the means was assumed to be 20%, therefore 20 patients per group are required, for a total of 60 patients. To these patients, the dropout percentage of 10% must be added, so the total is 70 patients.

T0 - BASELINE The first dental visit and the treatment plan will be carried out by Prof. Marco Dolci. The periodontal visit with the registration of the indices and the full-rx will be carried out by Prof. Marco Dolci.

Clinical indixes

* Bleeding On Probing - BOP, percentage value on 6 sites for each tooth
* Pocket Probing Depth - PPD on 6 sites for each tooth
* Clinical Attachment Loss - CAL on intraoral radiographs of pathological sites
* Plaque Index - PI, rated from 0 to 4 for each site
* Percentage of pathological sites out of total sites. The recording of BOP, PPD, PI will be carried out through periodontal probing using the PCP-15 UNC periodontal probe (HuFriedi) in a completely atraumatic and non-invasive manner.

The operational session will be organized as follows:

* Supragingival instrumentation with piezoelectric ultrasonic scaler handpiece;
* BPA microbiological test (Bacterial Periodontal Assessment - Biomolecular Diagnostic, Via Nicola Porpora, 550144 - Florence) through sampling of the gingival crevicular fluid with a thin cone of sterile paper with a diameter of 0.3 mm positioned in the pocket for 60 seconds, in an atraumatic and non-traumatic manner invasive. After sampling, the cones will be inserted into a single test tube;
* Subgingival instrumentation of periodontal pockets using Gracey curettes. The treatment is to be considered as Full Mouth Treatment (FMT). The samples will be transported to the laboratory located on the third floor of Building A, taken into custody by Prof. Marco Dolci and stored at + 4° C until the arrival of the dedicated courier.

The same Biomolecular Diagnostic company will take care of collecting the samples via dedicated biological courier and will carry out the PCR analyzes in its laboratories.

At the end of the analyses, a copy of a unique identification code will be sent to the Experimenters so that they can access the report.

Placement of the patient in the test, positive and negative control groups

TEST: home oral hygiene 2/day with soft bristle toothbrush + standard fluoride toothpaste + probiotic in buccal sachet to be consumed once a day until the quarterly check-up.

POSITIVE CONTROL: home oral hygiene 2/day with soft bristle toothbrush + standard fluoride toothpaste + industrial placebo in buccal sachet to be consumed once a day until the quarterly check-up.

NEGATIVE CONTROL: home oral hygiene 2/day with soft bristle toothbrush + standard fluoride toothpaste.

The products (test and placebo) will be delivered to the patient at the end of the session in order to cover 3 months of administration.

T1 - AFTER 3 MONTHS FROM T0

* Recording of periodontal indices.
* Microbiological samples.

Randomization The treatment that is due to the individual patient is kept in sequentially numbered, opaque and sealed envelopes (SNOSE Sequentially Numbered, Opaque, Sealed Envelopes). The products used for both the test and the controls will be supplied in anonymous tubes so that neither the patient nor the investigator will be aware of them.

Statistical analysis Proper statistical analysiswill be perfomed by the trusted statistical group.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the absence of other systemic pathologies reported in the medical history
* smokers and non-smokers, non-drinkers,
* subjects in the absence of previous or current administration of other sources of probiotics,
* subjects capable of providing informed consent.

Exclusion Criteria:

* Subjects with a history of systemic diseases (diabetes, autoimmune diseases, inflammatory bowel diseases, neurodegenerative diseases),
* drinkers,
* subjects who take or have taken probiotics in the last 3 months,
* subjects unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of clinical periodontal indexes | From enrollement to the end of treatment at 3 months.
  Evaluation of clinical periodontal indexes, such as: bleeding on probing (BOP), periodontal pocket depth (PPD), clinical attachment level (CAL), plaque index (PI), total number of pathological sites in %.

SECONDARY OUTCOMES:
Reduction of periodontal pathogen bacteria amount. | From enrollement to the end of treatment at 3 months.
  Evaluation of the amount of periodontal pathogen bacteria such as: A. actinomycetemcomitans, P. gingivalis, P. intermedia and F. nucleatum

CONTACTS AND LOCATIONS:
Overall Officials: Marco Dolci, MD DDS PHD, Principal Investigator — University G. d'Annunzio of Chieti
Locations (1):
- University G. d'Annunzio, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No
A decision regarding IPD sharing has not been made yet because a dedicated website is not available at the momente.

REFERENCES:
- [Background] Iwasaki K, Maeda K, Hidaka K, Nemoto K, Hirose Y, Deguchi S. Daily Intake of Heat-killed Lactobacillus plantarum L-137 Decreases the Probing Depth in Patients Undergoing Supportive Periodontal Therapy. Oral Health Prev Dent. 2016;14(3):207-14. doi: 10.3290/j.ohpd.a36099. PMID 27175447
- [Background] Sulijaya B, Takahashi N, Yamazaki K. Lactobacillus-Derived Bioactive Metabolites for the Regulation of Periodontal Health: Evidences to Clinical Setting. Molecules. 2020 Apr 29;25(9):2088. doi: 10.3390/molecules25092088. PMID 32365716
- [Background] Etebarian A, Sheshpari T, Kabir K, Sadeghi H, Moradi A, Hafedi A. Oral Lactobacillus species and their probiotic capabilities in patients with periodontitis and periodontally healthy individuals. Clin Exp Dent Res. 2023 Oct;9(5):746-756. doi: 10.1002/cre2.740. Epub 2023 Apr 20. PMID 37078410
- [Background] Pudgar P, Povsic K, Cuk K, Seme K, Petelin M, Gaspersic R. Probiotic strains of Lactobacillus brevis and Lactobacillus plantarum as adjunct to non-surgical periodontal therapy: 3-month results of a randomized controlled clinical trial. Clin Oral Investig. 2021 Mar;25(3):1411-1422. doi: 10.1007/s00784-020-03449-4. Epub 2020 Jul 14. PMID 32666349
- [Background] Mendi A, Kose S, Uckan D, Akca G, Yilmaz D, Aral L, Gultekin SE, Eroglu T, Kilic E, Uckan S. Lactobacillus rhamnosus could inhibit Porphyromonas gingivalis derived CXCL8 attenuation. J Appl Oral Sci. 2016 Jan-Feb;24(1):67-75. doi: 10.1590/1678-775720150145. PMID 27008259
- [Background] Gatej SM, Marino V, Bright R, Fitzsimmons TR, Gully N, Zilm P, Gibson RJ, Edwards S, Bartold PM. Probiotic Lactobacillus rhamnosus GG prevents alveolar bone loss in a mouse model of experimental periodontitis. J Clin Periodontol. 2018 Feb;45(2):204-212. doi: 10.1111/jcpe.12838. Epub 2017 Dec 11. PMID 29121411
- [Background] Morales A, Carvajal P, Silva N, Hernandez M, Godoy C, Rodriguez G, Cabello R, Garcia-Sesnich J, Hoare A, Diaz PI, Gamonal J. Clinical Effects of Lactobacillus rhamnosus in Non-Surgical Treatment of Chronic Periodontitis: A Randomized Placebo-Controlled Trial With 1-Year Follow-Up. J Periodontol. 2016 Aug;87(8):944-52. doi: 10.1902/jop.2016.150665. Epub 2016 Mar 4. PMID 26944407
- [Background] Fu J, Jia L, Wu L, Jiang Y, Zhao R, Du J, Guo L, Zhang C, Xu J, Liu Y. Lactobacillus rhamnosus inhibits osteoclast differentiation by suppressing the TLR2/NF-kappaB pathway. Oral Dis. 2024 May;30(4):2373-2386. doi: 10.1111/odi.14712. Epub 2023 Aug 21. PMID 37602540
- [Background] Routier A, Blaizot A, Agossa K, Dubar M. What do we know about the mechanisms of action of probiotics on factors involved in the pathogenesis of periodontitis? A scoping review of in vitro studies. Arch Oral Biol. 2021 Sep;129:105196. doi: 10.1016/j.archoralbio.2021.105196. Epub 2021 Jun 10. PMID 34153538
- [Background] Nguyen T, Brody H, Radaic A, Kapila Y. Probiotics for periodontal health-Current molecular findings. Periodontol 2000. 2021 Oct;87(1):254-267. doi: 10.1111/prd.12382. PMID 34463979
- [Background] Morales A, Gandolfo A, Bravo J, Carvajal P, Silva N, Godoy C, Garcia-Sesnich J, Hoare A, Diaz P, Gamonal J. Microbiological and clinical effects of probiotics and antibiotics on nonsurgical treatment of chronic periodontitis: a randomized placebo- controlled trial with 9-month follow-up. J Appl Oral Sci. 2018 Jan 18;26:e20170075. doi: 10.1590/1678-7757-2017-0075. PMID 29364340
- [Background] Teughels W, Durukan A, Ozcelik O, Pauwels M, Quirynen M, Haytac MC. Clinical and microbiological effects of Lactobacillus reuteri probiotics in the treatment of chronic periodontitis: a randomized placebo-controlled study. J Clin Periodontol. 2013 Nov;40(11):1025-35. doi: 10.1111/jcpe.12155. Epub 2013 Sep 15. PMID 24164569
- [Background] Furlaneto F, Ishikawa KH, Messora MR, Mayer MPA. Probiotics During the Therapeutic Management of Periodontitis. Adv Exp Med Biol. 2022;1373:353-375. doi: 10.1007/978-3-030-96881-6_19. PMID 35612808
- [Background] Gruner D, Paris S, Schwendicke F. Probiotics for managing caries and periodontitis: Systematic review and meta-analysis. J Dent. 2016 May;48:16-25. doi: 10.1016/j.jdent.2016.03.002. Epub 2016 Mar 8. PMID 26965080
- [Background] Lee Y, Yoon Y, Choi KH. Probiotics-Mediated Bioconversion and Periodontitis. Food Sci Anim Resour. 2021 Nov;41(6):905-922. doi: 10.5851/kosfa.2021.e57. Epub 2021 Nov 1. PMID 34796320
- [Background] Bustamante M, Oomah BD, Mosi-Roa Y, Rubilar M, Burgos-Diaz C. Probiotics as an Adjunct Therapy for the Treatment of Halitosis, Dental Caries and Periodontitis. Probiotics Antimicrob Proteins. 2020 Jun;12(2):325-334. doi: 10.1007/s12602-019-9521-4. PMID 30729452
- [Background] Sanz M, Ceriello A, Buysschaert M, Chapple I, Demmer RT, Graziani F, Herrera D, Jepsen S, Lione L, Madianos P, Mathur M, Montanya E, Shapira L, Tonetti M, Vegh D. Scientific evidence on the links between periodontal diseases and diabetes: Consensus report and guidelines of the joint workshop on periodontal diseases and diabetes by the International diabetes Federation and the European Federation of Periodontology. Diabetes Res Clin Pract. 2018 Mar;137:231-241. doi: 10.1016/j.diabres.2017.12.001. Epub 2017 Dec 5. PMID 29208508
- See also: New Classification of periodontal and peri-implant diseases — https://www.efp.org/fileadmin/uploads/efp/Documents/Campaigns/New_Classification/Guidance_Notes/report-02.pdf